CLINICAL TRIAL: NCT06421636
Title: A PHASE 2, TWO-PART, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY TO EVALUATE THE EFFICACY, SAFETY, AND TOLERABILITY OF SUBCUTANEOUSLY ADMINISTERED REGN7999 (AN INHIBITOR OF TMPRSS6) IN PARTICIPANTS WITH IRON OVERLOAD DUE TO NON-TRANSFUSION DEPENDENT β-THALASSEMIA
Brief Title: A Study to Test the Safety, Tolerability, and Efficacy of an Antibody, REGN7999, Injected Under the Skin for the Treatment of Iron Overload in Adult Participants With Non-Transfusion Dependent β-thalassemia, Using MRI Scans to Measure Iron Levels in the Body
Acronym: FERVENT-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7999-BThal-2350; 2023-508604-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non-Transfusion Dependent Beta-Thalassemia (NTDT)
Keywords: Beta-Thalassemia; Resultant Iron Overload (IOL)
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A High Dose (Experimental): Randomized 2:2:1
  Interventions: Drug: REGN7999
- Part A Low Dose (Experimental): Randomized 2:2:1
  Interventions: Drug: REGN7999
- Part A Placebo (Placebo Comparator): Randomized 2:2:1
  Interventions: Drug: Placebo
- Part B High Dose (Experimental): Randomized 2:2:1
  Interventions: Drug: REGN7999
- Part B Low Dose (Experimental): Randomized 2:2:1
  Interventions: Drug: REGN7999
- Part B Placebo (Placebo Comparator): Randomized 2:2:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN7999 — Administered subcutaneous (SC)
  Arms: Part A High Dose; Part A Low Dose; Part B High Dose; Part B Low Dose
Drug: Placebo — Administered SC
  Arms: Part A Placebo; Part B Placebo

SUMMARY:
This study is researching an experimental drug called REGN7999 (called "study drug"). The study is focused on patients with non-transfusion dependent beta-thalassemia. The aim of the study is to see how safe and effective the study drug is.

The study is looking at several other research questions, including:

* Whether the study drug lowers extra iron levels in the body
* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of NTDT as described in the protocol
2. IOL, defined as LIC ≥ 5 mg Fe/g DW as measured by R2* MRI at screening
3. Serum ferritin ≥ 300 ng/mL as described in the protocol

Key Exclusion Criteria:

1. Hemoglobin ≤ 8 g/dL at screening
2. Any RBC transfusion within 12 weeks of visit 3
3. For Part A only: Any Iron Chelation Therapy (ICT) use in approximately 12 weeks prior to screening as described in the protocol
4. For Part B only: If on ICT, any change in ICT dose in approximately 12 weeks prior to screening as described in the protocol
5. Any use of luspatercept or mitapivat in 6 months prior to screening as described in the protocol
6. Absolute contraindication to MRI
7. Diagnosis of cirrhosis of the liver
8. Diagnosis of Chronic kidney disease (CKD) stage 4 or higher

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-01-24 (Estimated); Study Completion 2028-01-24 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Liver Iron Concentration (LIC) by R2* Magnetic Resonance Imaging (MRI) | At week 24
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Up to week 72
Severity of TEAEs | Up to week 72

SECONDARY OUTCOMES:
Achievement of ≥20% reduction from baseline in LIC by R2* MRI | Through week 52
Change from baseline in hemoglobin | To week 24
Change from baseline in LIC by R2* MRI | At week 52
Percent change from baseline in LIC by R2* MRI | To week 24 and week 52
Achievement of ≥20% reduction from baseline in LIC by R2* MRI | Through week 24
Change in hemoglobin over time | Up to week 56
Achievement of ≥1.5 g/dL increase in hemoglobin for two consecutive assessments in the absence of Red Blood Cell (RBC) transfusions | Baseline to week 56
Number of RBC transfusions required | Baseline to week 72
Achievement of transfusion independence | Baseline to week 72
Change in RBC counts over time | Baseline to week 56
Concentrations of REGN7999 in serum over time | Up to week 56
Incidence of Anti-Drug Antibody (ADA) to REGN7999 over time | Up to week 56
Magnitude of ADA to REGN7999 over time | Up to week 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (25):
- Weill Cornell Medicine, New York, New York, United States
- Georgia (2):
  - K Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Medinvest Institute of Hematology and Transfusiology Limited, Tbilisi
- Greece (3):
  - Children's Hospital Agia Sophia, Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - University Hospital of Ioannina, Ioannina
- India (7):
  - Hemato-Oncology Clinic Ahmedabad PVT. LTD., Ahmedabad, Gujarat
  - Nirmal Hospital Pvt. Ltd - Surat, Surat, Gujarat
  - Amrita Institute of Medical Sciences and Research Centre (AIMS), Kochi, Kerala
  - K J Somaiya Super Specialty Hospital & Research Centre, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - JK Lon Hospital, Jaipur, Rajasthan
- Day Hospital Thalassemia and Haemoglobinopathies (DHTE); A.O.U S.Anna, Ferrara, Italy
- Malaysia (4):
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Ampang, Ampang, Selangor
  - Hospital Tunku Ampuan Besar Tuanku Aishah Rohani (HPKK UKM), Kuala Lumpur
- Thailand (5):
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Chulalongkorn University, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- United Kingdom (2):
  - University College London Hospitals NHS Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/